CLINICAL TRIAL: NCT03576014
Title: A Prospective, Open, Dose-escalation, Multi-center, Phase 1 Trial to Evaluate Tolerability and Safety of Intramuscularly Administered BD03, a DNA Vaccine for Prevention of CMV and BKV Reactivation in Kidney Transplant Recipient
Brief Title: Evaluate Tolerability and Safety of BD03 for Prevention of CMV and BKV Reactivation in Kidney Transplant Recipient
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SL VAXiGEN (Industry)
Collaborators: SL BIGEN (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BD03_KT_P1
Record Dates: First submitted 2018-05-25; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Cytomegalovirus Infections; Preventation of Cytomegalovirus Reactivation; BK Virus Infection; Preventation of BK Virus Reactivation
Keywords: CMV; BKV; CMV Reactivation; BKV Reactivation; DNA Vaccine; Kidney transplant; Cytomegalovirus; BK virus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD03 (Experimental): This study will be comprised of 3+3 dose escalation design with three dose levels, 0.6mg (cohort1), 2mg(cohort2), 6mg(cohort3).
  Decision to increase dose will be guided by occurrence of DLT (dose limiting toxicity) evaluated 1week after the second injection (5weeks after first injection)
  Interventions: Biological: BD03

INTERVENTIONS:
Biological: BD03 — BD03 is to be administered intramuscularly 6 weeks and 2 weeks prior to kidney transplant and 2~4 weeks after the transplant.

SUMMARY:
This study is a phase I, open-label study to determine recommended phase 2 dose (RP2D) for the BD03 vaccination in kidney transplant recipients. The recommended dose will be selected based on the safety and tolerability profiles observed.

DETAILED DESCRIPTION:
It is reported that CMV and BKV infection and/or reactivations are associated with mortality and morbidity of kidney transplant recipient, and occurrence of PyVAN in kidney transplant recipients.

BD03 is a DNA vaccine that consists of 3 plasmid DNAs encoding CMV antigens, BKV antigens and genetic adjuvant. It is expected to express antigen specific T-cell immune response, and ultimately prevent activation of both viruses. Plasmid DNA that encode CMV and BKV antigens are fused with tPA and Flt-3L to promote antigen specific immune response.

Patient scheduled to receive kidney transplant from living donor are enrolled in this study. Eligible subjects will receive BD03 intramuscularly by electroporator three times on 6 weeks and 2 weeks prior to kidney transplant and 2~4 weeks after the transplant.

This study will be comprised of 3+3 dose escalation scheme and starting dose is 0.6mg and dose will be increased to 2mg and 6mg.

Occurrence of dose limiting toxicities observed until 1 week after second injection (1week before kidney transplant) will guide whether to increase a dose.

After third injection of BD03, follow up visits are done for 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 19
* Body Mass Index ≤ 35
* Weight ≥ 40kg

Exclusion Criteria:

* CMV IgG seronegative patient
* Patient scheduled for retransplant of kidney
* Patient known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
* Patient expected to receive T-cell depleting agents or rituximab
* Patient with history of splenectomy
* Patient with CMV related disease or shows active CMV infection or who has been treated with CMV related disease or CMV infection within 3 months from consent date.
* Patient expected to undergo CMV prophylaxis using anti-virals or immunoglobulins.
* Patient who has hypersensitivity to BD03 or components of BD03.
* Patient with history of epilepsy or seizure with the last 2 years
* Patients with pre-excitation syndrome or any other disease who would be considered ineligible for electroporation injection.
* Patient with blood coagulation disorder who would be considered ineligible for electroporation injection
* Patient with injection site thickness greater than 40mm
* Patient with artificial implant near injection site
* Pregnant or breast-feeding female patient
* Female subject or partner of male subject with child bearing potential and who has not agreed to sexual abstinence
* Patient who has participated in any other clinical trial within 30 days
* Patient who has any clinically meaningful disease investigator's judgement to prevent participating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-07-24 (Estimated)

PRIMARY OUTCOMES:
Tolerability as measured by dose-limiting toxicities (DLTs) | 5 weeks
  An event will be considered a DLT if the event is reasonably related to study treatment during the 5weeks of treatment, and meets the following criteria: Any Grade 3 or greater toxicity per CTCAE 4.03 that would be considered dose-limiting except for those associated with kidney failure, Grade 3 or greater Creatine kinase increase that is not accompanied with Rhabdomyolysis, and any other Grade3 or greater toxicity that exists before participation of this study.

SECONDARY OUTCOMES:
Proportion of subjects whose Spot Forming Units per unit PBMC are tripled compared to base line measurements and subjects whose Spot Forming Units of each antigen in 10^6 PBMC are greater than 50. | Up to 30 weeks post-dose
  To evaluate the immunogenicity of BD03. ELISPOT assay of specific T cell responses to CMV and BKV antigens.
Antibody response to CMV gB antigen | Up to 30 weeks post-dose
  To investigate antibody level measured by Enzyme-Linked ImmunoSorbent Assay(ELISA)
Antibody response to BKV VP1 antigen | Up to 30 weeks post-dose
  To investigate antibody level measured by Enzyme-Linked ImmunoSorbent Assay(ELISA)
Change of CMV and BKV plasma viral load over time | Up to 30 weeks post-dose
  To investigate change of CMV and BKV plasma viral load over time

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical center, Seoul
  - Seoul St.Mary's Hospital, Seoul

REFERENCES:
- [Background] Hirsch HH, Randhawa P; AST Infectious Diseases Community of Practice. BK polyomavirus in solid organ transplantation. Am J Transplant. 2013 Mar;13 Suppl 4:179-88. doi: 10.1111/ajt.12110. PMID 23465010
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597